CLINICAL TRIAL: NCT02863770
Title: Prospective Controlled Trial of Contrast Enhanced Endoscopic Ultrasound for Evaluation of Pancreas Lesions
Brief Title: Contrast EUS of the Pancreas
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, James Buxbaum, Associate Professor of Clinical Medicine, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HS-15-00784
Record Dates: First submitted 2016-08-01; First posted 2016-08-11 (Estimated); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Pancreatic Neoplasms; Pancreatitis; Pancreatic Cyst
Keywords: endosonography
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatitis; Pancreatic Cyst

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Contrast EUS (Experimental): Undergoing EUS for pancreatic indication (cyst, pancreatitis, mass)
  Interventions: Other: EUS enhanced with contrast to evaluate pancreas

INTERVENTIONS:
Other: EUS enhanced with contrast to evaluate pancreas — Patients will receive intravenous contrast during EUS to assess whether it increases diagnostic yield of the examination

SUMMARY:
RATIONALE: Endoscopic Ultrasound (EUS) is the leading method to evaluate the pancreas but there may be difficulty characterizing small lesions, tumors which are not adenocarcinomas and neoplasia in the setting of pancreatitis.

INTERVENTION: The innovation in this project will be the addition of intravenous contrast to standard EUS examination if the pancreas.

PURPOSE: The aim is to determine if contrast enhances the ability of EUS to accurately diagnose lesions and target biopsies, and to define the quantitative features of this method.

STUDY POPULATION:The population will include patients with pancreas cysts, masses, and inflammation presenting for EUS as part of standard clinical care.

METHODOLOGY: This will be a prospective tandem trial involving conventional EUS, followed by EUS with contrast, followed by subsequent quantitative processing of contrast EUS imaging.

ENDOINTS:Study endpoints will include the yield contrast EUS to evaluate pancreas cysts, masses, and inflammation. The impact of contrast EUS to better target the FNA of the chosen lesion will be assessed. Intra and interobserver variability will be assessed by comparing conventional EUS and contrast EUS of each case in a random order (intraobserver agreement) and among a group of blinded endosonographers (interobserver agreement).

DETAILED DESCRIPTION:
AIM Early detection of pancreas cancer and precursors lesions improves survival. The investigators aim is to gauge whether quantitative contrast endoscopic ultrasound (EUS) improves the evaluation of pancreas tumors and precursors lesions including cysts.

DESIGN The study will be a prospective tandem contrast EUS trial. All EUS will be performed as part of standard clinical care.

Conventional EUS Standard EUS will first be performed using the 180 series linear array echoendoscope (Olympus, Center Valley, PA). The alpha-10 image processor (Aloka America, Wallingford, CT) in B mode will be used to acquire images. A research coordinator will help to record key parameters. Thirty second cine clips of conventional EUS images will be captured to compare with contrast EUS clips and enable intra and interobserver variability comparison.

Contrast Administration Definity contrast will be activated by 45 seconds of agitation (VialMix, Lantheus, North Billerica, MA) and injected through the intravenous peripheral line which is placed to administer fluids. The investigators will administer a bolus dose of 10microliter (microL)/kg within 30-60 seconds followed by 10ml of saline flush. Up to 2 bolus injections will be administered during each case and doppler sonography will be used between them to induce microbubble destruction.

Contrast EUS: Following contrast administration prospective assessment will be performed using the Olympus endoscope and images processed using the Alpha 10 system. Harmonic detection conversion software installed on the alpha 10 processor to enable detection. Core parameters for comparison to conventional EUS will be captured prospectively.

Quantitative Processing: For each bolus 30 seconds of cine imaging will be captured for post processing and for comparison with conventional EUS imaging (intra and interobserver variability). Images of the lesion (5mm x 5mm region) and adjacent normal tissue (5mm x 5mm) regions will be captured to facilitate quantitative assessment. Quantitative analytic software will then be used to generate time intensity curves and associated values including peak intensity (PI), time to peak (TTP), wash-in-slope (WIS), rise time (RT), mean transit time (MTT), and time from peak to one-half (TPH).

DRUG/DEVICE INFORMATION

Definity: Definity is an intravenous contrast agent. It is comprised of 1.1-3.3um micropheres containing perflutren (octafluoropropane) which is cleared by respiration.

The gas is encapsulated lipid shells which are metabolized to free fatty acids and hepatically cleared.

The Olympus 180 linear echoendoscope will be used in all procedures which are being done for standard clinical indications. The Aloka SSD-Alpha 10-Processor will be used for image capture. Post EUS quantitative processing will be performed using QLAB quantification software (Philips Healthcare, Bothel, WA).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing endoscopic ultrasound for standard pancreatic indications.
* Patients must have unexplained pancreatitis, pancreas mass(es), or pancreatic cystic lesions (>1cm or worrisome features on imaging).

Exclusion Criteria:

* Patients <18 years of age, pregnant women, and lactating mothers will be excluded. Subjects with unstable ischemic disease will be excluded. Additionally, those with known or suspected right-to-left, bi-directional, or transient right-to-left cardiac shunts will be excluded given theoretical (though clinically insignificant) risk of embolization.
* Patients with an allergy to Definity will be excluded.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-07; Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
The yield of EUS versus contrast EUS to diagnose pancreas cystic lesions, mass lesion, and origin of pancreatitis. | 6 months
  The endoscopist will perform conventional EUS and classify the lesion as described below, this will be recorded by the research assistant prior to contrast EUS. Contrast will then be administered and the classification of contrast EUS recorded in real time. The gold standard to calculate the yields of the modality will be on pathology and clinical diagnosis at three and six months. Additionally we will assess whether contrast impacted assessment of size and diagnosis.

SECONDARY OUTCOMES:
Targeting of FINE NEEDLE ASPIRATION (FNA) of pancreas lesions. | 6 months
  A) The decision to perform a FINE NEEDLE ASPIRATION of the lesion will be based solely on the standard EUS exam. After making the decision to perform the FNA contrast EUS will be performed. We will assess the degree to whether contrast administration helped to better target the FNA of the chosen lesion
Quantitative Parameters of Pancreas Lesions | 6 months
  Quantitative parameters of pancreas mass lesions will be performed by comparing the quantitative parameters post processing of adenocarcinoma, neuroendocrine and other lesion, and chronic pancreatitis. The final diagnosis will be based on pathology and 3 and 6 month follow up. Comparison variables will include time to peak (SECONDS), rise time (SECONDS), mean transit time (SECONDS), and time from peak to one-half (SECONDS).

CONTACTS AND LOCATIONS:
Locations (1):
- Los Angeles County Hospital, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Napoleon B, Alvarez-Sanchez MV, Gincoul R, Pujol B, Lefort C, Lepilliez V, Labadie M, Souquet JC, Queneau PE, Scoazec JY, Chayvialle JA, Ponchon T. Contrast-enhanced harmonic endoscopic ultrasound in solid lesions of the pancreas: results of a pilot study. Endoscopy. 2010 Jul;42(7):564-70. doi: 10.1055/s-0030-1255537. Epub 2010 Jun 30. PMID 20593334
- [Background] Kitano M, Kudo M, Yamao K, Takagi T, Sakamoto H, Komaki T, Kamata K, Imai H, Chiba Y, Okada M, Murakami T, Takeyama Y. Characterization of small solid tumors in the pancreas: the value of contrast-enhanced harmonic endoscopic ultrasonography. Am J Gastroenterol. 2012 Feb;107(2):303-10. doi: 10.1038/ajg.2011.354. Epub 2011 Oct 18. PMID 22008892
- [Background] Saftoiu A, Vilmann P, Dietrich CF, Iglesias-Garcia J, Hocke M, Seicean A, Ignee A, Hassan H, Streba CT, Ioncica AM, Gheonea DI, Ciurea T. Quantitative contrast-enhanced harmonic EUS in differential diagnosis of focal pancreatic masses (with videos). Gastrointest Endosc. 2015 Jul;82(1):59-69. doi: 10.1016/j.gie.2014.11.040. Epub 2015 Mar 16. PMID 25792386
- [Background] King KG, Gulati M, Malhi H, Hwang D, Gill IS, Cheng PM, Grant EG, Duddalwar VA. Quantitative assessment of solid renal masses by contrast-enhanced ultrasound with time-intensity curves: how we do it. Abdom Imaging. 2015 Oct;40(7):2461-71. doi: 10.1007/s00261-015-0468-y. PMID 26036794